CLINICAL TRIAL: NCT00956163
Title: F-18 NaF PET for Detection of Bone Metastases in Men With Prostate Cancer: Exploratory Study
Brief Title: Whole Body Fluorine F 18 Sodium Fluoride PET/CT Scan and Whole Body MRI in Finding Bone Metastases in Patients With Prostate Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NCI-2011-02972; NCI-2011-02972 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000666327; MGH-09364; 09-364 (Other: Massachusetts General Hospital Cancer Center); 8336 (Other: CTEP); P30CA006516 (NIH); N01CM37120 (NIH)
Record Dates: First submitted 2009-08-07; First posted 2009-08-11 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2013-12

CONDITIONS: Bone Metastases; Recurrent Prostate Cancer; Stage I Prostate Cancer; Stage IIA Prostate Cancer; Stage IIB Prostate Cancer; Stage III Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Technetium Tc 99m Medronate

ARMS (1):
- Diagnostic (fluorine F 18 sodium fluoride PET) (Experimental): Patients undergo technetium Tc 99m methylene diphosphonate bone scan, fluorine F 18 sodium fluoride PET/CT scan, and whole-body MRI for the detection of bone metastases. Patients with discordant imaging results (negative bone scan and positive PET/CT scan and/or MRI) undergo additional imaging at 6, 12, 18, and 24 months.
  Interventions: Procedure: magnetic resonance imaging; Radiation: fluorine F 18 sodium fluoride; Procedure: positron emission tomography; Procedure: computed tomography; Radiation: technetium Tc 99m methylene diphosphonate; Other: laboratory biomarker analysis

INTERVENTIONS:
Procedure: magnetic resonance imaging — Undergo whole-body MRI
  Other Names: MRI; NMR imaging; NMRI; nuclear magnetic resonance imaging
Radiation: fluorine F 18 sodium fluoride — Undergo fluorine F 18 sodium fluoride PET/CT scan
  Other Names: 18 F-NaF; F-18 NaF
Procedure: positron emission tomography — Undergo fluorine F 18 sodium fluoride PET/CT scan
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed
Procedure: computed tomography — Undergo fluorine F 18 sodium fluoride PET/CT scan
  Other Names: tomography, computed
Radiation: technetium Tc 99m methylene diphosphonate — Undergo technetium Tc 99m methylene diphosphonate bone scan
  Other Names: 99mTc-MDP; TechneScan MDP; technetium Tc 99m medronate
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase 0 trial studies whole body fluorine F 18 sodium fluoride positron emission tomography (PET)/computed tomography (CT) scan and whole body magnetic resonance imaging (MRI) in finding bone metastases in patients with prostate cancer. Diagnostic procedures, such as whole body fluorine F 18 sodium fluoride PET/CT scan and whole body MRI, may help find and diagnose bone metastases.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the sensitivity and specificity of whole-body fluorine F 18 sodium fluoride PET/CT scan in detecting bone metastases in patients with high-risk prostate cancer using bone scan as the reference standard.

II. To evaluate the sensitivity and specificity of whole-body MRI in detecting bone metastases in patients with high-risk prostate cancer using bone scan as the reference standard.

OUTLINE:

Patients undergo technetium Tc 99m methylene diphosphonate bone scan, fluorine F 18 sodium fluoride PET/CT scan, and whole-body MRI for the detection of bone metastases. Patients with discordant imaging results (negative bone scan and positive PET/CT scan and/or MRI) undergo additional imaging at 6, 12, 18, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Any ethnic group
* Pathologically proven prostate cancer with high risk for bone metastases
* Rising prostate-specific antigen (PSA) despite androgen deprivation therapy (ADT), PSA > 10 ng/mL
* Ability to understand and the willingness to sign a written combined Health Insurance Portability and Accountability Act (HIPAA) and informed consent document
* Patients Eastern Cooperative Oncology Group (ECOG) performance is =< 1

Exclusion Criteria:

* Patients may not receive any other investigational therapeutic agents from within 7 days prior to study drug administration through 7 days following study drug administration
* Patients with known contraindications to MR imaging such as presence of MRI incompatible devices such as pacemakers and certain aneurysm clips, severe claustrophobia, or any other condition which would preclude proximity to a strong magnetic field; this exclusion is a standard of practice
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements; patients in this category are excluded to reduce medical risk to their safety and to avoid confounding variables in regard to the possibility of adverse events
* Patient is unable to tolerate or has a lifer threatening allergy to the radiopharmaceutical used for bone scan or 18F-fluoride PET

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-03; Primary Completion 2011-01 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Uptake of fluorine F 18 sodium fluoride on PET/CT scan | Up to 24 months
  Determine if increased uptake of 18F-fluoride on PET/CT scan is directly correlated to the metastatic tumor burden within the bones using bone scan as the reference standard.
Incidence of focal MRI abnormality | Up to 24 months
  Determine if focal MRI abnormality is directly correlated to the metastatic tumor burden within the bones using bone scan as the reference standard.

CONTACTS AND LOCATIONS:
Overall Officials: Mukesh Harisinghani, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States